CLINICAL TRIAL: NCT03988738
Title: Social Media-based Intervention to Promote Repeat Blood Donation Among First-time Blood Donors in a Peruvian Blood Bank: Randomized Controlled Trial
Brief Title: Promoting Repeat Blood Donation Through Social Media Among First-time Donors in a Peruvian Blood Bank
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Principal Investigator, Joel Gustavo Rondón Rodríguez, Researcher, Universidad Peruana Cayetano Heredia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 103806
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Blood Donors
Keywords: Blood Donors; Social Media; Blood Donation; Facebook; WhatsApp

STUDY DESIGN:
Intervention Model Description: Donors will be randomly assigned to one of two groups using complete block randomization until a total of 212 participants are recruited: 106 in the intervention group and 106 in the control group.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive messages regarding blood donation promotion and campaigns through social media once or twice a week for six months.
  Interventions: Other: Social Media Publications
- Control (Sham Comparator): Participants will receive a message regarding blood donation at the beginning of the study through social media. After four months they will receive another message including information about upcoming blood donation campaigns.
  Interventions: Other: Social Media Publications

INTERVENTIONS:
Other: Social Media Publications — Messages will be elaborated prior to participant enrollment. Messages will be evaluated by three experts.

SUMMARY:
Blood donations are an important need worldwide. In Peru, only 10% of donations are voluntary, of which only a quarter are repeat donors. Repeat donations are crucial to maintaining a safe and adequate blood supply.

Social media presents a unique opportunity to promote blood donation, because of its increasing use and its prior successes in promoting positive health-related behaviors .

The present study aims to develop and evaluate a social media intervention - Facebook and WhatsApp - to improve communication and promote repeat blood donations in voluntary first-time donors attending donation campaigns organized by the Hospital Nacional Cayetano Heredia (HCH).

DETAILED DESCRIPTION:
Main Objective:

To evaluate the effect of social media in the promotion of repeat blood donation among first-time blood donors in a Peruvian blood bank.

Study design:

A randomized control trial will be conducted over a 6-month period, and will compare the rate of repeat blood donation who amongst first-time donors who received promotional messages through social media and those who did not.

Population:

Voluntary first-time blood donors who attend blood donation campaigns organized by the blood bank of the Hospital Nacional Cayetano Heredia (HCH), Lima - Peru.

Sample:

A sample of 105 participants per group was calculated, with a significance of 95% and a power of 80%, to show a difference of 20% in recurrence rate of blood donation between the two groups.

Group assignment:

Participant selection will occur at blood donation campaigns organized by the HCH blood bank. If inclusion and exclusion criteria are met, donors will be invited to participate in the study. After accepting and signing the informed consent form, donors will be randomly assigned to one of two groups using complete block randomization until a total of 212 participants are recruited: 106 in the intervention group and 106 in the control group. All participants will receive an introductory message through social media confirming their participation in the study.

Ethical considerations:

Written informed consent will be requested from participants. Data confidentiality will be maintained. Personal identifiers will be stored in a separate database, which will be password protected and accessible only to the research team.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary first-time Blood Donor
* Eligible to donate blood again
* Facebook or WhatsApp user

Exclusion Criteria:

* Denial to participate in the study
* Refusal to be contacted by social media

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-01-25 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Repeat Blood donation rate | 6 months
  Rate of repeat blood donation will be assessed in both groups after intervention.

SECONDARY OUTCOMES:
Time interval between blood donations | 6 months
  Time interval between blood donations will be evaluated in both groups.
Readiness to Change | 6 months
  Apply Transtheoretical Model of Change to assess first-time donors´ readiness to change.

CONTACTS AND LOCATIONS:
Overall Officials: Joel G Rondon Rodriguez, MD, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (1):
- Hospital Nacional Cayetano Heredia Blood Bank, San Martín de Porres, Lima region, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George PE, Vidal J, Garcia PJ. An Analysis of and Recommendations for the Peruvian Blood Collection and Transfusion System. J Epidemiol Public Health Rev. 2016 May;1(3):10.16966/2471-8211.119. doi: 10.16966/2471-8211.119. Epub 2016 Apr 22. PMID 27761524
- [Background] Househ M. The use of social media in healthcare: organizational, clinical, and patient perspectives. Stud Health Technol Inform. 2013;183:244-8. PMID 23388291
- [Background] Schmunis GA, Cruz JR. Safety of the blood supply in Latin America. Clin Microbiol Rev. 2005 Jan;18(1):12-29. doi: 10.1128/CMR.18.1.12-29.2005. PMID 15653816
- [Background] Hagg E, Dahinten VS, Currie LM. The emerging use of social media for health-related purposes in low and middle-income countries: A scoping review. Int J Med Inform. 2018 Jul;115:92-105. doi: 10.1016/j.ijmedinf.2018.04.010. Epub 2018 Apr 26. PMID 29779724
- [Background] Burditt C, Robbins ML, Paiva A, Velicer WF, Koblin B, Kessler D. Motivation for blood donation among African Americans: developing measures for stage of change, decisional balance, and self-efficacy constructs. J Behav Med. 2009 Oct;32(5):429-42. doi: 10.1007/s10865-009-9214-7. Epub 2009 Apr 14. PMID 19365718
- [Background] Amoyal NR, Robbins ML, Paiva AL, Burditt C, Kessler D, Shaz BH. Measuring the processes of change for increasing blood donation in black adults. Transfusion. 2013 Jun;53(6):1280-90. doi: 10.1111/j.1537-2995.2012.03864.x. Epub 2012 Aug 28. PMID 22928841
- [Background] World Health Organization, International Federation of Red Cross and Red Crescent Societies. Towards 100% voluntary blood donation: A global framework for action [Internet]. Geneva: WHO; 2010 [cited 2019 Jan 29]. Available from: https://www.who.int/bloodsafety/publications/9789241599696_eng.pdf
- [Background] Frye V, Duffy L, France JL, Kessler DA, Rebosa M, Shaz BH, Carlson BW, France CR. The Development of a Social Networking-Based Relatedness Intervention Among Young, First-Time Blood Donors: Pilot Study. JMIR Public Health Surveill. 2018 Apr 26;4(2):e44. doi: 10.2196/publichealth.8972. PMID 29699961
- [Background] Dirección General de Donaciones Trasplantes y Banco de Sangre. Peruvian National Plan for Voluntary Blood Donor Promotion 2018 - 2021 [Internet]. Lima: Peru Ministry of Health; 2018 p. 16. Available from: ftp://ftp2.minsa.gob.pe/normaslegales/2018/Resolucion_Ministerial_672-2018-MINSA.pdf